CLINICAL TRIAL: NCT02073968
Title: PET-Adjusted IMRT for NSCLC Trial (PAINT)
Brief Title: PET-Adjusted Intensity Modulated Radiation Therapy and Combination Chemotherapy in Treating Patients With Stage II-IV Non-small Cell Lung Cancer
Acronym: PAINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-252; NCI-2014-00216 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-252 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Recurrent Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes; Magnetic Resonance Spectroscopy; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (PET-adjusted IMRT, carboplatin, paclitaxel) (Experimental): RADIOTHERAPY: Patients undergo PET-adjusted IMRT or proton beam radiation therapy five days a week for 5 weeks.
  CONCURRENT CHEMOTHERAPY: Patients receive carboplatin IV over 3 hours and paclitaxel IV over 1 hour once weekly for 6 weeks beginning week 1 of thoracic radiotherapy.
  CONSOLIDATION CHEMOTHERAPY: Beginning approximately 4-6 weeks after the completion of all radiation therapy and when esophagitis and chemotherapy-induced neuropathy are grade 1 or less, ANC > 1500, and platelet count > 100,000, patients may receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment may repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity at the discretion of the treating physicians.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Radiation: Intensity-Modulated Radiation Therapy; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Radiation: Proton Beam Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo PET-adjusted IMRT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: Intensity-Modulated Radiation Therapy — Undergo PET-adjusted IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo PET-adjusted IMRT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy

SUMMARY:
This phase II trial studies how well intensity modulated radiation therapy adjusted by positron emission tomography (PET) scanning together with combination chemotherapy works in treating patients with stage II-IV non-small cell lung cancer (NSCLC). Radiation therapy uses high energy x rays to kill tumor cells. In intensity-modulated radiotherapy, multiple beam angles and dozens of beam segments are used to deliver highly conformal radiation therapy. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving PET-adjusted IMRT together with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy (based on post-treatment PET findings) of dose-painted intensity-modulated radiotherapy (IMRT) with concurrent chemotherapy for locally-advanced non-small cell lung cancer (LA-NSCLC).

SECONDARY OBJECTIVES:

I. To estimate the efficacy (based on clinical endpoints including locoregional control [LRC], disease-free survival [DFS], and overall survival [OS]) of dose-painted IMRT with concurrent chemotherapy for LA-NSCLC.

II. To evaluate the safety of dose-painted IMRT with concurrent and adjuvant chemotherapy for LA-NSCLC.

III. To evaluate the utility of post-treatment PET/computed tomography (CT) imaging as a predictor of clinical outcomes following treatment with this novel approach.

IV. To explore, in a preliminary manner, whether metabolomic markers in the blood and urine prior to and during the course of treatment are associated with treatment response, clinical endpoints, and treatment-related adverse events such as radiation pneumonitis.

OUTLINE:

RADIATION THERAPY: Patients undergo PET-adjusted IMRT or proton beam radiation therapy five days a week for 5 weeks.

CONCURRENT CHEMOTHERAPY: Patients receive carboplatin intravenously (IV) over 3 hours and paclitaxel IV over 1 hour once weekly for 5 weeks beginning week 1 of thoracic radiotherapy.

CONSOLIDATION CHEMOTHERAPY: Beginning approximately 4-6 weeks after the completion of all radiation therapy and when esophagitis and chemotherapy-induced neuropathy are grade 1 or less, absolute neutrophil count (ANC) > 1500, and platelet count > 100,000, patients may receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment may repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity at the discretion of the treating physicians.

After completion of study treatment, patients are followed up at 12-16 weeks, 19 weeks, every 3 months for 2 years, and then every 6 months for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of NSCLC with any of the following stages (according to the American Joint Committee on Cancer [AJCC] Staging Manual, 7th edition):

  * Stage IIIA or IIIB
  * Stage II NSCLC with medical contraindication to curative surgical resection
  * Stage IV disease with solitary brain metastasis that has been treated radically (eg: with surgical resection or stereotactic radiosurgery) and thoracic disease that would be classified as stage II-III
* Appropriate diagnostic/staging workup, including:

  * Complete history and physical examination
  * Whole body PET/computed tomography (CT) scan within 42 days prior to study entry demonstrating hypermetabolic pulmonary lesion(s) and/or thoracic lymph node(s), with a maximum standardized uptake volume (SUV) > 6 for at least one lesion; if PET/CT was obtained more than 42 days prior to study entry and is not repeated, CT scan of the chest within 28 days prior to study entry demonstrating stable disease is required
  * Magnetic resonance imaging (MRI) of the brain or CT scan of the head with contrast within 42 days prior to study entry
  * Biopsy confirmation of suspected metastatic disease identified by PET/CT is recommended
  * Pulmonary function tests (PFTs) within 6 weeks of study entry are highly recommended but not required
* No prior chemotherapy or thoracic radiotherapy for lung cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500 cells/ul
* Platelets >= 100,000 cells/ul
* Hemoglobin >= 9.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 9.0 g/dl is acceptable)
* Total bilirubin < 3.0 times the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x the ULN
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance >= 50 ml/min (by Cockroft-Gault formula)
* Women of childbearing potential must:

  * Have a negative serum or urine pregnancy test within 72 hours prior to the start of study therapy
  * Agree to utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study therapy is completed
  * Be advised of the importance of avoiding pregnancy during trial participation and the potential risks of an unintentional pregnancy
* All patients must sign study specific informed consent prior to study entry

Exclusion Criteria:

* Pleural or pericardial effusion

  * A patient with pleural effusion may be enrolled the effusion is sampled by thoracentesis and cytology is negative or the effusion is seen on axial imaging but not on chest x-ray and deemed too small to tap under CT or ultrasound guidance
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
* Women who

  * Are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study therapy
  * Have a positive pregnancy test at baseline
  * Are pregnant or breastfeeding
* Poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL) despite attempts to improve glucose control by fasting duration and adjustment of medications; patients with diabetes will preferably be scheduled for PET/CT imaging in the morning, and instructions for fasting and use of medications will be provided in consultation with the patients' primary physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel): RADIOTHERAPY: Patients undergo PET-adjusted IMRT five days a week for 5 weeks.
  CONCURRENT CHEMOTHERAPY: Patients receive carboplatin paclitaxel weekly for 5 weeks during thoracic radiotherapy.
  OPTIONAL CONSOLIDATION CHEMOTHERAPY: Beginning approximately 4-6 weeks after the completion of radiotherapy, subjects may receive up to 3 cycles of consolidation carboplatin and paclitaxel.
Period: Overall Study
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 35 subjects received study therapy. 30 subjects underwent post-treatment PET/CT and were eligible for analysis with respect to the primary study endpoint.
Groups:
- Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel): RADIOTHERAPY: Patients undergo PET-adjusted IMRT five days a week for 5 weeks.
  CONCURRENT CHEMOTHERAPY: Patients receive carboplatin IV over 3 hours and paclitaxel IV over 1 hour once weekly for 6 weeks beginning week 1 of thoracic radiotherapy.
  CONSOLIDATION CHEMOTHERAPY: Beginning approximately 4-6 weeks after the completion of all radiation therapy and when esophagitis and chemotherapy-induced neuropathy are grade 1 or less, ANC > 1500, and platelet count > 100,000, patients may receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment may repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity at the discretion of the treating physicians.
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo PET-adjusted IMRT
  Paclitaxel: Given IV
  Positron Emission Tomography: Undergo PET-adjusted IMRT
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Full Range); unit: years] | 68 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Response of All Pulmonary Lesions and Thoracic Lymph Nodes
Description: Favorable response will be defined as having maximum SUV less than 6.0 on post-treatment PET/CT.
Time Frame: Up to 16 weeks after completion of radiation therapy
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel): RADIOTHERAPY: Patients undergo PET-adjusted IMRT or proton beam radiation therapy five days a week for 5 weeks.
  CONCURRENT CHEMOTHERAPY: Patients receive carboplatin IV over 3 hours and paclitaxel IV over 1 hour once weekly for 6 weeks beginning week 1 of thoracic radiotherapy.
  CONSOLIDATION CHEMOTHERAPY: Beginning approximately 4-6 weeks after the completion of all radiation therapy patients may receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment may repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity at the discretion of the treating physicians.
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo PET-adjusted IMRT
  Paclitaxel: Given IV
  Positron Emission Tomography: Undergo PET-adjusted IMRT
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 30
Participants | 24

2. Secondary Outcome: Incidence of Grade >= 2 Radiation-induced Lung Toxicity, Scored Using Common Terminology Criteria for Adverse Events (CTCAE), Version (v.) 4
Description: Incidence of grade >= 2 radiation-induced lung toxicity, scored using Common Terminology Criteria for Adverse Events (CTCAE), version (v.) 4, will be presented as frequency and percentages.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel): RADIOTHERAPY: Patients undergo PET-adjusted IMRT or proton beam radiation therapy five days a week for 5 weeks.
  CONCURRENT CHEMOTHERAPY: Patients receive carboplatin IV over 3 hours and paclitaxel IV over 1 hour once weekly for 6 weeks beginning week 1 of thoracic radiotherapy.
  CONSOLIDATION CHEMOTHERAPY: Beginning approximately 4-6 weeks after the completion of all radiation therapy and when esophagitis and chemotherapy-induced neuropathy are grade 1 or less, ANC > 1500, and platelet count > 100,000, patients may receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment may repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity at the discretion of the treating physicians.
  Carboplatin: Given IV
  Computed Tomography: Undergo PET-adjusted IMRT
  Intensity-Modulated Radiation Therapy: Undergo PET-adjusted IMRT
  Paclitaxel: Given IV
  Positron Emission Tomography: Undergo PET-adjusted IMRT
  Proton Beam Radiation Therapy: Undergo proton beam radiation therapy
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 35
Participants | 7

3. Secondary Outcome: Incidence of Grade >= 3 Treatment-related Toxicity, Scored Using CTCAE, v. 4
Description: Incidence of grade >= 3 treatment-related toxicity, scored using CTCAE, v. 4, will be presented as frequency and percentages.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 35
Participants | 30

4. Secondary Outcome: Locoregional Progression-free Survival Assessed Using the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  Kaplan-Meier survival plots will be produced. The survival probabilities will be presented.
Time Frame: From study registration to date of local or regional disease progression or death, censored at the date of data collection, assessed at 1 year
Measure: Number; unit: percentage with LRPFS at 1 year
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 35
percentage with LRPFS at 1 year | 50

5. Secondary Outcome: Lung Cancer Cause-specific Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  A patient will be considered to have died from lung cancer if he or she had evidence of disease progression at any site and no direct evidence of other cause of death. Kaplan-Meier survival plots will be produced.
Time Frame: From study registration to death directly from lung cancer, censored at the date of data collection, up to a maximum of 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 35
months | 28 [28 to 28]

6. Secondary Outcome: Overall Survival
Description: Kaplan-Meier survival plots will be produced. The survival probabilities will be presented. Log-rank testing will be used to compare the survival probabilities between categorical predictors. A Cox regression model will be used to estimate the hazard rates for overall survival among the predictor variables.
Time Frame: From study registration to death, censored at the date of data collection, assessed at 1 year
Measure: Number; unit: percentage of patients alive at 1 year
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 35
percentage of patients alive at 1 year | 74

7. Secondary Outcome: Progression-free Survival Assessed Using the RECIST Criteria
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  Kaplan-Meier survival plots will be produced. The survival probabilities will be presented. Log-rank testing will be used to compare the survival probabilities between categorical predictors. A Cox regression model will be used to estimate the hazard rates for progression free survival among the predictor variables.
Time Frame: From study registration to date of disease progression or death, censored at the date of data collection, assessed at 1 year
Measure: Number; unit: percentage of patients w/ PFS at 1 year
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 35
percentage of patients w/ PFS at 1 year | 26

ADVERSE EVENTS:
Time Frame: Median follow-up time is 5.5 months for the entire cohort and 23.8 months for surviving patients.
Description: Adverse events were scored using Common Terminology Criteria for Adverse Events version 4.0 at each study visit. Adverse events occurring within 90 days of radiation therapy completion were categorized as acute toxicities, and subsequent adverse events were categorized as late toxicities.
Groups:
- Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel): RADIOTHERAPY: Patients undergo PET-adjusted IMRT or proton beam radiation therapy five days a week for 5 weeks.
  CONCURRENT CHEMOTHERAPY: Patients receive carboplatin IV over 3 hours and paclitaxel IV over 1 hour once weekly for 6 weeks beginning week 1 of thoracic radiotherapy.
  CONSOLIDATION CHEMOTHERAPY: Beginning approximately 4-6 weeks after the completion of all radiation therapy, patients may receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment may repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity at the discretion of the treating physicians.
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo PET-adjusted IMRT
  Paclitaxel: Given IV
  Positron Emission Tomography: Undergo PET-adjusted IMRT
Arm/Group | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 11/35
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel) (N=35)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (PET-adjusted IMRT, Carboplatin, Paclitaxel) (N=35)
Anorexia (Gastrointestinal disorders) | 14 (14)
Constipation (Gastrointestinal disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (25)
Dermatitis (Skin and subcutaneous tissue disorders) | 19 (19)
Dysphagia (Gastrointestinal disorders) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT02073968/Prot_SAP_000.pdf